CLINICAL TRIAL: NCT04421547
Title: Phase III Randomized Control Case Study of Letrozole in Women With Heavily Pretreated Ovarian Cancer (MITO32)
Brief Title: Efficacy of Letrozole in Recurrent Ovarian Cancer
Acronym: MITO32
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Logistical problems impacting the speed of enrolment
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, MARCHETTI CLAUDIA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MITO32
Record Dates: First submitted 2020-05-15; First posted 2020-06-09 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Epithelial Ovarian Cancer
Keywords: epithelial ovarian cancer; Letrozole
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Letrozole

STUDY DESIGN:
Intervention Model Description: This is a two arms, prospective, open-label multi center randomized phase III study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letrozole (Experimental): Letrozole 1 tablet (2,5 mg) orally once a day
  Interventions: Drug: Letrozole 2.5mg
- Standard Chemotherapy (Active Comparator): Either Paclitaxel 80 mg/m2 as a 1-h infusion, on days 1,8,15,22 every 28 days or Pegylated Liposomal Doxorubicin (PLD) 40 mg/m2 given every 4 weeks or Topotecan 4mg/m2 IV on days 1,8,15 every 4 weeks or Gemcitabine 1000 mg/m2 IV over 30 min on days 1,8,15 every 28 days.
  Interventions: Drug: Standard single agent chemotherapy

INTERVENTIONS:
Drug: Letrozole 2.5mg — This study will investigate the role of Letrozole in patients affected by heavily pretreated platinum resistant ovarian cancer, compared to standard treatment.
  Arms: Letrozole
Drug: Standard single agent chemotherapy — Either Paclitaxel 80 mg/m2 as a 1-h infusion, on days 1,8,15,22 every 28 days or Pegylated Liposomal Doxorubicin (PLD) 40 mg/m2 given every 4 weeks or Topotecan 4mg/m2 IV on days 1,8,15 every 4 weeks or Gemcitabine 1000 mg/m2 IV over 30 min on days 1,8,15 every 28 days.
  Arms: Standard Chemotherapy

SUMMARY:
Randomized phase III multicenter study investigating the role of letrozole in heavily pretreated recurrent ovarian cancer.

DETAILED DESCRIPTION:
This is a randomized, open-label, phase III, multicenter, global study evaluating the efficacy and safety of Letrozole in heavily pretreated recurrent ovarian cancer patients in comparison to physician' choice chemotherapy.

Subjects who meet all the inclusion criteria and none of the exclusion criteria will be randomized in a 1:1 ratio to one of the two arms, as follow:

Arm A: Letrozole 1 tablet (2,5 mg) orally once a day in 28-day cycles Arm B: Pegylated Liposomal Doxorubicin 40 mg/m2 d1q28 or Topotecan 4 mg/m2 d1,8,15q28 or Gemcitabine 1000 mg/m2 d1,8,15q28 or Paclitaxel 80 mg/m2 d1,8,15q28 In case of objective response and acceptable toxicity, no maximum number of cycles of treatment is defined.

The aim of the study is to assess the activity of Letrozole in women with recurrent epithelial ovarian cancer, heavily pretreated.

ELIGIBILITY:
Inclusion Criteria:

* Female of 18 years of age or older
* Histologically or cytologically documented invasive epithelial ovarian cancer, primary peritoneal carcinoma, or fallopian tube cancer
* Platinum resistant or refractory disease (patients who did not respond to last platinumbased therapy or with last relapse occurred < 6 months from the last dose of platinum) or patients not amenable of platinum treatment
* >3 previous chemotherapy lines
* ECOG performance status 0 -2
* Measurable and evaluable disease according to RECIST criteria confirmed by radiological imaging: at least one lesion of ≥ 1.0 cm for non-lymph nodes or ≥ 1.5 cm in short-axis diameter for lymph nodes at CT scan (Subjects with isolated rising CA-125 without radiologically visible disease are excluded)
* Left Ventricular Ejection Fraction (LVEF) ≥ institutional lower limit normal
* Estimated life expectancy ≥ 16 weeks
* Adequate functions evidenced by:

  * Hemoglobin ³10.0 g/dl
  * Absolute neutrophil count ³1.5 x 109/L
  * White blood cells >3x109/L
  * Platelet >100 x109/L
  * AST and ALT £ 2.5 x Upper limit of normal, unless liver metastasis, in which case AST and ALT < or = 5 x Upper limit of normal will be accepted
  * Bilirubin ≤ 1.5 times the upper limit of normal (ULN)
  * Estimated glomerular filtration ³ 60mL/min using the Cockcroft-Gault equation.
* Patient able to comply with the treatment
* Evidence of not pregnancy status as documented by a negative beta-human chorionic gonadotropin (ß-hCG) test
* Not breastfeeding women
* Patients with child-bearing potential using (or willing to use) effective contraception during treatment and 3 months ahead unless they are postmenopausal (at least 12 months consecutive amenorrhea, in the appropriate age group and without other known or suspected cause), or have been sterilized surgically.
* Comprehension and signature of the informed consent

Exclusion Criteria:

* Subjects with borderline ovarian cancer
* Subject with low malignant potential tumors
* Less than 3 lines of previous therapies
* Platinum sensitive disease (last relapse occurred > 6 months from the last dose of platinum)
* Less than 4 weeks from last dose of therapy with any investigational agent, or chemotherapy
* History of another neoplastic disease (except basal cell carcinoma or cervical carcinoma in situ adequately treated) unless in remission for 3 years or longer
* Breastfeeding women
* Pregnant women
* Prior therapy with letrozole.
* Severe osteoporosis documented by BMD (Bone Mineral Density) T-score ≤ -2.5 with existing fragility fracture(s)
* Patients with a known hypersensitivity to Paclitaxel , PLD, Topotecan, Gemcitabine or Letrozole or any case of severe toxicity related to them. Also Patients with a known hypersensitivity to any of the ingredients or excipients of the IMPs (e.g. macrogolglycerol ricinoleate (polyoxyl castor oil), ethanol, anhydrous, citric acid, anhydrous, sodium chloride hydrochloric acid, mannitol, sodium acetate, sodium hydroxide, tartaric acid, lactose monohydrate, maize starch, hypromellose Type 2910, cellulose microcrystalline, sodium starch glycolate type A, colloidal anhydrous silica, magnesium stearate, hypromellose 6 cp E464, titanium dioxide E171, Iron oxide yellow E172, Macrogol 400, talc E553b)
* Prior resistance to Paclitaxel, PLD, Topotecan, Gemcitabine
* Patients with active hepatic disease (HCV or HBV infections), hepatic severe impairment or cirrhosis
* Bowel obstruction, sub-occlusive disease, prior gastrectomy, symptomatic brain metastases.
* Myocardial infarct within six months before enrolment , NYHA Class II or worse heart failure, unstable angina, serious cardiac arrhythmia or cardiac arrhythmia requiring treatment.
* Any serious concomitant illness requiring treatment
* Pre-existing peripheral neuropathy > CTCAE Grade 2.
* Concomitant use of strong CYP3A4 inhibitors (e.g. ketoconazole, itraconazole, voriconazole, ritonavir, clarithromycin, and telithromycin) or strong CYP2A6 inhibitors (e.g. methoxsalen) because they may increase exposure to letrozole.
* Concomitant use of inducers of CYP3A4 (e.g. phenytoin, rifampicin, carbamazepine, phenobarbital, and St. John's Wort) which may reduce exposure to letrozole.
* Concomitant use of medicinal products with a narrow therapeutic index that are substrates for CYP2C19 (e.g. phenytoin, clopidrogel) that may have their systemic serum concentrations altered by letrozole.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patient alive at 12 months | 30 months
  Evaluate the difference in terms of proportion of survivals at 12 months between the two arms.

SECONDARY OUTCOMES:
PFS | 30 months
  Progression Free Survival
OS | 30 months
  Overall Survival
ORR | 30 months
  Objective Response Rate (according to RECIST criteria version 1.1)
TPST | 30 months
  Time from randomization to the start of the primary subsequent therapy
TSST | 30 months
  Time from randomization to the start of the secondary subsequent therapy
Toxicity profile evaluated according to NCI-CTCAE version 5.0 | 30 months
  Toxicity profile (evaluated according to NCI-CTCAE version 5.0)
QoL | 30 months
  Quality of Life (evaluated by EORTC QLQ-C30/ QLQ-OV28 questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Marchetti, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- DH Tumori Femminili, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Banerjee S, Kaye SB, Ashworth A. Making the best of PARP inhibitors in ovarian cancer. Nat Rev Clin Oncol. 2010 Sep;7(9):508-19. doi: 10.1038/nrclinonc.2010.116. Epub 2010 Aug 10. PMID 20700108
- [Background] Banerjee S, Kaye SB. New strategies in the treatment of ovarian cancer: current clinical perspectives and future potential. Clin Cancer Res. 2013 Mar 1;19(5):961-8. doi: 10.1158/1078-0432.CCR-12-2243. Epub 2013 Jan 10. PMID 23307860
- [Background] Gore ME, Fryatt I, Wiltshaw E, Dawson T. Treatment of relapsed carcinoma of the ovary with cisplatin or carboplatin following initial treatment with these compounds. Gynecol Oncol. 1990 Feb;36(2):207-11. doi: 10.1016/0090-8258(90)90174-j. PMID 2404837
- [Background] Markman M, Rothman R, Hakes T, Reichman B, Hoskins W, Rubin S, Jones W, Almadrones L, Lewis JL Jr. Second-line platinum therapy in patients with ovarian cancer previously treated with cisplatin. J Clin Oncol. 1991 Mar;9(3):389-93. doi: 10.1200/JCO.1991.9.3.389. PMID 1999708
- [Background] Buda A, Floriani I, Rossi R, Colombo N, Torri V, Conte PF, Fossati R, Ravaioli A, Mangioni C. Randomised controlled trial comparing single agent paclitaxel vs epidoxorubicin plus paclitaxel in patients with advanced ovarian cancer in early progression after platinum-based chemotherapy: an Italian Collaborative Study from the Mario Negri Institute, Milan, G.O.N.O. (Gruppo Oncologico Nord Ovest) group and I.O.R. (Istituto Oncologico Romagnolo) group. Br J Cancer. 2004 Jun 1;90(11):2112-7. doi: 10.1038/sj.bjc.6601787. PMID 15150623
- [Background] Sehouli J, Stengel D, Oskay-Oezcelik G, Zeimet AG, Sommer H, Klare P, Stauch M, Paulenz A, Camara O, Keil E, Lichtenegger W. Nonplatinum topotecan combinations versus topotecan alone for recurrent ovarian cancer: results of a phase III study of the North-Eastern German Society of Gynecological Oncology Ovarian Cancer Study Group. J Clin Oncol. 2008 Jul 1;26(19):3176-82. doi: 10.1200/JCO.2007.15.1258. PMID 18591555
- [Background] ten Bokkel Huinink W, Gore M, Carmichael J, Gordon A, Malfetano J, Hudson I, Broom C, Scarabelli C, Davidson N, Spanczynski M, Bolis G, Malmstrom H, Coleman R, Fields SC, Heron JF. Topotecan versus paclitaxel for the treatment of recurrent epithelial ovarian cancer. J Clin Oncol. 1997 Jun;15(6):2183-93. doi: 10.1200/JCO.1997.15.6.2183. PMID 9196130
- [Background] Gordon AN, Fleagle JT, Guthrie D, Parkin DE, Gore ME, Lacave AJ. Recurrent epithelial ovarian carcinoma: a randomized phase III study of pegylated liposomal doxorubicin versus topotecan. J Clin Oncol. 2001 Jul 15;19(14):3312-22. doi: 10.1200/JCO.2001.19.14.3312. PMID 11454878
- [Background] Mutch DG, Orlando M, Goss T, Teneriello MG, Gordon AN, McMeekin SD, Wang Y, Scribner DR Jr, Marciniack M, Naumann RW, Secord AA. Randomized phase III trial of gemcitabine compared with pegylated liposomal doxorubicin in patients with platinum-resistant ovarian cancer. J Clin Oncol. 2007 Jul 1;25(19):2811-8. doi: 10.1200/JCO.2006.09.6735. PMID 17602086
- [Background] Vergote I, Finkler NJ, Hall JB, Melnyk O, Edwards RP, Jones M, Keck JG, Meng L, Brown GL, Rankin EM, Burke JJ, Boccia RV, Runowicz CD, Rose PG. Randomized phase III study of canfosfamide in combination with pegylated liposomal doxorubicin compared with pegylated liposomal doxorubicin alone in platinum-resistant ovarian cancer. Int J Gynecol Cancer. 2010 Jul;20(5):772-80. doi: 10.1111/igc.0b013e3181daaf59. PMID 20973267
- [Background] Pujade-Lauraine E, Hilpert F, Weber B, Reuss A, Poveda A, Kristensen G, Sorio R, Vergote I, Witteveen P, Bamias A, Pereira D, Wimberger P, Oaknin A, Mirza MR, Follana P, Bollag D, Ray-Coquard I. Bevacizumab combined with chemotherapy for platinum-resistant recurrent ovarian cancer: The AURELIA open-label randomized phase III trial. J Clin Oncol. 2014 May 1;32(13):1302-8. doi: 10.1200/JCO.2013.51.4489. Epub 2014 Mar 17. PMID 24637997
- [Background] Lakusta CM, Atkinson MJ, Robinson JW, Nation J, Taenzer PA, Campo MG. Quality of life in ovarian cancer patients receiving chemotherapy. Gynecol Oncol. 2001 Jun;81(3):490-5. doi: 10.1006/gyno.2001.6199. PMID 11371144
- [Background] Demers LM, Melby JC, Wilson TE, Lipton A, Harvey HA, Santen RJ. The effects of CGS 16949A, an aromatase inhibitor on adrenal mineralocorticoid biosynthesis. J Clin Endocrinol Metab. 1990 Apr;70(4):1162-6. PMID 2156889
- [Background] Lipton A, Demers LM, Harvey HA, Kambic KB, Grossberg H, Brady C, Adlercruetz H, Trunet PF, Santen RJ. Letrozole (CGS 20267). A phase I study of a new potent oral aromatase inhibitor of breast cancer. Cancer. 1995 Apr 15;75(8):2132-8. doi: 10.1002/1097-0142(19950415)75:83.0.co;2-u. PMID 7697604
- [Background] El Ouagari K, Karnon J, Delea T, Talbot W, Brandman J. Cost-effectiveness of letrozole in the extended adjuvant treatment of women with early breast cancer. Breast Cancer Res Treat. 2007 Jan;101(1):37-49. doi: 10.1007/s10549-006-9262-4. Epub 2006 Jul 4. PMID 16821085
- [Background] Sioufi A, Gauducheau N, Pineau V, Marfil F, Jaouen A, Cardot JM, Godbillon J, Czendlik C, Howald H, Pfister C, Vreeland F. Absolute bioavailability of letrozole in healthy postmenopausal women. Biopharm Drug Dispos. 1997 Dec;18(9):779-89. doi: 10.1002/(sici)1099-081x(199712)18:93.0.co;2-5. PMID 9429742
- [Background] Sioufi A, Sandrenan N, Godbillon J, Trunet P, Czendlik C, Howald H, Pfister C, Ezzet F. Comparative bioavailability of letrozole under fed and fasting conditions in 12 healthy subjects after a 2.5 mg single oral administration. Biopharm Drug Dispos. 1997 Aug;18(6):489-97. doi: 10.1002/(sici)1099-081x(199708)18:63.0.co;2-p. PMID 9267682
- [Background] Dave N, Gudelsky GA, Desai PB. The pharmacokinetics of letrozole in brain and brain tumor in rats with orthotopically implanted C6 glioma, assessed using intracerebral microdialysis. Cancer Chemother Pharmacol. 2013 Aug;72(2):349-57. doi: 10.1007/s00280-013-2205-y. Epub 2013 Jun 9. PMID 23748921
- [Background] Lamb HM, Adkins JC. Letrozole. A review of its use in postmenopausal women with advanced breast cancer. Drugs. 1998 Dec;56(6):1125-40. doi: 10.2165/00003495-199856060-00020. PMID 9878997
- [Background] Goss PE, Ingle JN, Martino S, Robert NJ, Muss HB, Piccart MJ, Castiglione M, Tu D, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Therasse P, Palmer MJ, Pater JL. A randomized trial of letrozole in postmenopausal women after five years of tamoxifen therapy for early-stage breast cancer. N Engl J Med. 2003 Nov 6;349(19):1793-802. doi: 10.1056/NEJMoa032312. Epub 2003 Oct 9. PMID 14551341
- [Background] Batra S, Iosif CS. Elevated concentrations of antiestrogen binding sites in membrane fractions of human ovarian tumors. Gynecol Oncol. 1996 Feb;60(2):228-32. doi: 10.1006/gyno.1996.0030. PMID 8631543
- [Background] Langdon SP, Gourley C, Gabra H, Stanley B. Endocrine therapy in epithelial ovarian cancer. Expert Rev Anticancer Ther. 2017 Feb;17(2):109-117. doi: 10.1080/14737140.2017.1272414. Epub 2016 Dec 24. PMID 27967255
- [Background] Slotman BJ, Rao BR. Ovarian cancer (review). Etiology, diagnosis, prognosis, surgery, radiotherapy, chemotherapy and endocrine therapy. Anticancer Res. 1988 May-Jun;8(3):417-34. PMID 3291746
- [Background] Langdon SP, Hawkes MM, Lawrie SS, Hawkins RA, Tesdale AL, Crew AJ, Miller WR, Smyth JF. Oestrogen receptor expression and the effects of oestrogen and tamoxifen on the growth of human ovarian carcinoma cell lines. Br J Cancer. 1990 Aug;62(2):213-6. doi: 10.1038/bjc.1990.263. PMID 2386737
- [Background] Langdon SP, Crew AJ, Ritchie AA, Muir M, Wakeling A, Smyth JF, Miller WR. Growth inhibition of oestrogen receptor-positive human ovarian carcinoma by anti-oestrogens in vitro and in a xenograft model. Eur J Cancer. 1994;30A(5):682-6. doi: 10.1016/0959-8049(94)90545-2. PMID 8080688
- [Background] O'Donnell AJ, Macleod KG, Burns DJ, Smyth JF, Langdon SP. Estrogen receptor-alpha mediates gene expression changes and growth response in ovarian cancer cells exposed to estrogen. Endocr Relat Cancer. 2005 Dec;12(4):851-66. doi: 10.1677/erc.1.01039. PMID 16322326
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Papadimitriou CA, Markaki S, Siapkaras J, Vlachos G, Efstathiou E, Grimani I, Hamilos G, Zorzou M, Dimopoulos MA. Hormonal therapy with letrozole for relapsed epithelial ovarian cancer. Long-term results of a phase II study. Oncology. 2004;66(2):112-7. doi: 10.1159/000077436. PMID 15138362
- [Background] Bowman A, Gabra H, Langdon SP, Lessells A, Stewart M, Young A, Smyth JF. CA125 response is associated with estrogen receptor expression in a phase II trial of letrozole in ovarian cancer: identification of an endocrine-sensitive subgroup. Clin Cancer Res. 2002 Jul;8(7):2233-9. PMID 12114425
- [Background] Markman M, Iseminger KA, Hatch KD, Creasman WT, Barnes W, Dubeshter B. Tamoxifen in platinum-refractory ovarian cancer: a Gynecologic Oncology Group Ancillary Report. Gynecol Oncol. 1996 Jul;62(1):4-6. doi: 10.1006/gyno.1996.0181. PMID 8690289
- [Background] Ferrandina G, Ludovisi M, Lorusso D, Pignata S, Breda E, Savarese A, Del Medico P, Scaltriti L, Katsaros D, Priolo D, Scambia G. Phase III trial of gemcitabine compared with pegylated liposomal doxorubicin in progressive or recurrent ovarian cancer. J Clin Oncol. 2008 Feb 20;26(6):890-6. doi: 10.1200/JCO.2007.13.6606. PMID 18281662
- [Background] Le T, Leis A, Pahwa P, Wright K, Ali K, Reeder B, Kinderchuck M, Ward K. Quality of life evaluations of caregivers of ovarian cancer patients during chemotherapy treatment. J Obstet Gynaecol Can. 2004 Jul;26(7):627-31. doi: 10.1016/s1701-2163(16)30609-0. PMID 15248931
- [Background] Stiggelbout AM, de Haes JC. Patient preference for cancer therapy: an overview of measurement approaches. J Clin Oncol. 2001 Jan 1;19(1):220-30. doi: 10.1200/JCO.2001.19.1.220. PMID 11134216